CLINICAL TRIAL: NCT03015428
Title: "Living Together With Dementia"_Creation and Validation of a Training Program for Family Caregivers of People With Dementia to Live at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Lia Sousa, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LTWD1
Record Dates: First submitted 2016-04-10; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Dementia
Keywords: Family caregivers; training programme; dementia
MeSH Terms: conditions — Dementia

ARMS (1):
- Psychoeducation (Experimental): Interventions:
  Give information Teach and train strategies
  Interventions: Other: psychoeducation

INTERVENTIONS:
Other: psychoeducation — Providing knowledge and skills development in family caregivers of people with dementia, through a structured psychoeducational programme

SUMMARY:
This study aims to experimentally evaluate the training program for family caregivers of people with dementia_"Living together with Dementia."

DETAILED DESCRIPTION:
This study will begin in March 2016, with the initial assessment of family caregivers of people with dementia.

These were recruited through hospital neurology clinic and must comply with a set of pre-established criteria.

It is expected a total of 20 participants in the study (10 in the experimental group and 10 in control group).

Interventions will take place over the months of March and April. The final evaluation is scheduled for late April and the follow up to July 2016.

an evaluation document itself for this study was built.

ELIGIBILITY:
Inclusion Criteria:

* Be primary caregiver of the person with dementia
* Be able to read and write
* Carers of peolpe with dementia in initial or moderate stage

Exclusion Criteria:

* The person with dementia have severe mental pathologies associated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Caregiver Overload Scale | 7 weeks
Carers Assessment Satisfaction Index | 7 weeks
Carers Assessment Difficulties Index | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lia Sousa, Master, Principal Investigator — Centro Hospitalar De São João, E.P.E.
Locations (1):
- CHSaoJoao, Porto, Portugal